CLINICAL TRIAL: NCT04430894
Title: A Phase II Study of Once Weekly Carfilzomib, Lenalidomide, Dexamethasone, and Isatuximab in Newly Diagnosed, Transplant-Eligible Multiple Myeloma
Brief Title: KRDI in Transplant-Eligible MM
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Amgen (Industry); Sanofi (Industry)
Responsible Party: Principal Investigator, Noopur Raje, Principal Investigator, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 19-568
Record Dates: First submitted 2020-06-11; First posted 2020-06-12 (Actual); Results first posted 2023-10-26 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; isatuximab; Lenalidomide; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Induction (Experimental): All participants will receive 4 cycles of induction therapy. Based on the recommendation of investigators, participants may or may not proceed to an autologous stem cell transplant (SCT) after cycles 1-4. Each cycle is 28 days in length (see dosing details below.)
  For patient undergoing upfront stem cell transplant (SCT): 4 cycles followed by stem cell collection, high-dose chemotherapy, and autologous SCT followed by 2 cycles (called consolidation).
  For patients deferring SCT following collection: 4 cycles followed by stem cell collection followed by 4 additional cycles.
  Carfilzomib: 56 mg/m2 IV on days 1, 8,15 Lenalidomide 25 mg orally (PO) on Days 1-21 Isatuximab: 10 mg/kg IV weekly for cycles 1-2 (days 1, 8, 15, 22), then every 2 weeks for cycles 3-6 (days 1 and 15), and monthly (day 1) thereafter Dexamethasone: 20 mg orally (PO) administered day of and day after carfilzomib and isatuximab (days 1, 2, 8, 9, 15, and 16; days 22 and 23 during cycles 1-2 only).
  Interventions: Drug: Carfilzomib; Drug: Isatuximab; Drug: Lenalidomide; Drug: Dexamethasone
- Maintenance-High Risk (Experimental): Only patients that have achieved a partial response (PR) or better after induction therapy with or without stem cell transplant will continue on to maintenance therapy. The treatment participants will receive for maintenance will be based on the biological features (or cytogenetics) of participants myeloma and categorized into two groups: Standard-risk and High Risk.
  High Risk: subjects with high risk cytogenetics (deletion (del 17, translocation (t)(4:14), t(14;16), t(14;20), 1q duplications) will receive the following study treatment for up to two years (24 28-day cycles) until progressive disease (PD) or unacceptable toxicity:
  Lenalidomide 10 mg orally (PO) Day 1-21 Carfilzomib 56 mg/m2 or last tolerated dose IV Days 1, 15 Isatuximab 10 mg/kg IV Day 1
  Interventions: Drug: Carfilzomib; Drug: Isatuximab; Drug: Lenalidomide; Drug: Dexamethasone
- Maintenance- Standard Risk (Experimental): Only patients that have achieved a partial response (PR) or better after induction therapy with or without stem cell transplant will continue on to maintenance therapy. The treatment participants will receive for maintenance will be based on the biological features (or cytogenetics) of participants myeloma and categorized into two groups: Standard-risk and High Risk.
  Standard Risk: subjects without high risk cytogenetics (deletion (del 17, translocation (t)(4:14), t(14;16), t(14;20), 1q duplications) will receive the following study treatment for up to two years (24 28-day cycles) until progressive disease (PD) or unacceptable toxicity:
  - Lenalidomide 10 mg orally (PO) Day 1-21
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Carfilzomib — * Induction: protocol determine dose,via IV on 3 days per cycle up to 8 cycles, dependent on Upfront Stem Transplant or Deferring Stem Cell Transplant determination
  * Maintenance: protocol determine dose,via IV on 2 days per cycle- Maintenance Cycle until progressive disease (PD) or unacceptable toxicity
  Other Names: Kyprolis
  Arms: Induction; Maintenance-High Risk
Drug: Isatuximab — * Induction: At predetermined dose, via IV up to 8 cycles, dependent on Upfront Stem Transplant or Deferring Stem Cell Transplant determination:
    -- Cycles 1 and 2 once per week, Cycles 3-4 every other week, Cycles 5 and 6 every other week, Cycles 7 and 8 once every 4 weeks.
  * Maintenance: At predetermined dose, via IV, once per cycle, Maintenance Cycle until progressive disease (PD) or unacceptable toxicity
  Other Names: Sarclisa
  Arms: Induction; Maintenance-High Risk
Drug: Lenalidomide — - Induction Predetermined Dose, oral, days 1-21 of up to 8 cycles, dependent on Upfront Stem Transplant or Deferring Stem Cell Transplant determination Maintenance: At predetermined dose, oral days 1-21 per cycle until progressive disease (PD) or unacceptable toxicity
  Other Names: REVLIMID
Drug: Dexamethasone — Induction: Predetermined dosage, oral, Predetermined times per cycle up to 8 cycles dependent on Upfront Stem Transplant or Deferring Stem Cell Transplant determination Maintenance: orally or IV will be administered as a preinfusion medication prior to isatuximab dosing
  Other Names: Decadron
  Arms: Induction; Maintenance-High Risk

SUMMARY:
This research study is testing the efficacy of an experimental drug combination for people with newly diagnosed multiple myeloma that are eligible for a stem cell transplant.

The names of the study drugs involved in this study are:

* Carfilzomib
* Isatuximab
* Lenalidomide
* Dexamethasone

DETAILED DESCRIPTION:
This is a phase II study to evaluate the efficacy of once weekly carfilzomib, lenalidomide, dexamethasone, and isatuximab (KRDI) in patients with newly diagnosed, transplant-eligible multiple myeloma. The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits. The study treatment portion of this study is comprised of an induction phase and a maintenance phase.

* Induction Phase :

  * All participants will receive the same study drugs (carfilzomib, isatuximab, lenalidomide, and dexamethasone) for up to 8 cycles. Each cycle is 28 days in length.
  * All participants will perform stem cell collection after 4 cycles of therapy. Based on the recommendation participants may or may not proceed to an autologous stem cell transplant (SCT) as part of induction therapy.
* Maintenance Phase: During maintenance, participants will receive the study treatment for up to two years after induction until progressive disease or unacceptable toxicity

It is expected that about 50 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational drug combination to learn whether the drug combination works in treating a specific disease.

"Investigational" means that the drug combination is being studied.

The U.S. Food and Drug Administration (FDA) has approved carfilzomib or isatuximab as a treatment for relapsed/refractory multiple myeloma.

The FDA has also approved lenalidomide and dexamethasone as a treatment option for transplant-eligible multiple myeloma.

However, the FDA has not approved the combination of isatuximab, carfilzomib, lenalidomide, and dexamethasone as an approved regimen. The combination is considered to be investigational for the treatment of individuals with newly diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age.
* Subject must have documented multiple myeloma satisfying the CRAB criteria and measurable disease defined as:

  * Monoclonal plasma cells in the bone marrow ≥10% or presence of a biopsy-proven Plasmacytoma.
  * Measurable disease as defined by any of the following:
  * IgG myeloma: Serum monoclonal paraprotein (M-protein) level ≥.5 g/dL or urine M-protein level ≥200 mg/24 hours; or
  * IgA, IgM, or IgD multiple myeloma: serum M-protein level ≥0.25 g/dL or urine M-protein level ≥200 mg/24 hours; or
  * Light chain multiple myeloma: Serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio.
  * Sixty percent or greater clonal plasma cells on bone marrow examination.
  * Serum involved / uninvolved free light chain ratio of 100 or greater, provided the absolute level of the involved free light chain is at least 100 mg/L (a patient's "involved" free light chain - either kappa or lambda - is the one that is above the normal reference range; the uninvolved light chain is the one that typically is in, or below, the normal range).
  * More than one focal lesion on magnetic resonance image (MRI) that is at least 5 mm or greater in size.
* Newly diagnosed and considered candidate for high-dose chemotherapy with stem cell transplant.
* Subject must have an Eastern Cooperative Oncology Group (ECOG) performance status score of 0, 1, or 2.
* Subject must have pretreatment clinical laboratory values meeting the following criteria during the Screening Phase:

  * hemoglobin ≥ 7.5 g/dL (≥ mmol/L; prior RBC transfusion or recombinant human erythropoietin use is permitted);
  * absolute neutrophil count ≥1.0 x 109/L (granulocyte colony stimulating factor [GCSF] use is permitted);
  * platelet count ≥70 x 109/L for subjects in whom <50% of bone marrow nucleated cells are plasma cells; otherwise platelet count >50 × 109/L (transfusions are not permitted to achieve this minimum platelet count)
  * aspartate aminotransferase (AST) ≤2.5 x upper limit of normal (ULN);
  * alanine aminotransferase (ALT) ≤2.5 x ULN;
  * total bilirubin ≤2.0 x ULN, except in subjects with congenital bilirubinemia, such as Gilbert syndrome (direct bilirubin ≤2.0 x ULN)
  * creatinine clearance ≥30 mL/min
  * corrected serum calcium ≤14 mg/dL (≤3.5 mmol/L); or free ionized calcium <6.5 mg/dL (<1.6 mmol/L).
* Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use 2 methods of reliable birth control simultaneously. This includes one highly effective form of contraception (tubal ligation, intrauterine device [IUD], hormonal [birth control pills, injections, hormonal patches, vaginal rings or implants] or partner's vasectomy) and one additional effective contraceptive method (male latex or synthetic condom, diaphragm, or cervical cap). Contraception must begin 4 weeks prior to dosing. Reliable contraception is indicated even where there has been a history of infertility, unless due to hysterectomy or bilateral oophorectomy.
* A man who is sexually active with a woman of childbearing potential must agree to use a latex or synthetic condom, even if they had a successful vasectomy. All men must also not donate sperm during the study, for 4 weeks after the last dose of lenalidomide, for 90 days after the last dose of carfilzomib, and for 4 months after the last dose of isatuximab.
* A woman of childbearing potential must have 2 negative serum or urine pregnancy tests at Screening, first within 10 to 14 days prior to dosing and the second within 24 hours prior to dosing.
* Each subject (or their legally acceptable representative) must sign an informed consent form (ICF) indicating that he or she understands the purpose of and procedures required for the study and are willing to participate in the study. Subject must be willing and able to adhere to the prohibitions and restrictions specified in this protocol, as referenced in the ICF.

Exclusion Criteria:

* Any potential subject who meets any of the following criteria will be excluded from participating in the study.
* Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, or smoldering multiple myeloma. Monoclonal gammopathy of undetermined significance is defined by presence of serum M-protein <3 g/dL; absence of lytic bone lesions, anemia, hypercalcemia, and renal insufficiency related to the M-protein; and (if determined) proportion of plasma cells in the bone marrow of 10% or less. Smoldering multiple myeloma is defined as asymptomatic MM with absence of related organ or tissue impairment end organ damage.
* Subject has a diagnosis of Waldenström's disease, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions
* Subject has prior or current systemic therapy or SCT for MM, with the exception of an emergency use of a short course (equivalent of dexamethasone 40 mg/day for a maximum 4 days) of corticosteroids before treatment.
* Subject has a history of malignancy (other than MM) within 5 years before the date of enrollment (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix, or malignancy that in the opinion of the investigator, with concurrence with the sponsor's medical monitor, is considered cured with minimal risk of recurrence within 5 years).
* Subject has had radiation therapy within 14 days of enrollment.
* Subject has had plasmapheresis within 28 days of enrollment.
* Subject is exhibiting clinical signs of meningeal involvement of MM.
* Subject has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume [FEV] in 1 second <60% of predicted normal), persistent asthma, or a history of asthma within the last 2 years (intermittent asthma is allowed). Subjects with known or suspected COPD or asthma must have a FEV1 test during screening.
* Subject is known to be seropositive for history of human immunodeficiency virus (HIV) or known to have active hepatitis B or hepatitis C.
* Subject has any concurrent medical or psychiatric condition or disease (eg, active systemic infection, uncontrolled diabetes, acute diffuse infiltrative pulmonary disease) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study.
* Subject has clinically significant cardiac disease, including:

  * myocardial infarction within 1 year before enrollment, or an unstable or uncontrolled disease/condition related to or affecting cardiac function (eg, unstable angina, congestive heart failure, New York Heart Association Class III-IV;
  * uncontrolled cardiac arrhythmia (National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4 Grade ≥2) or clinically significant ECG abnormalities;
  * screening 12-lead ECG showing a baseline QT interval as corrected by Fridericia's formula (QTcF) >470 msec.
  * uncontrolled hypertension
* Subject has known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to respective package inserts or IB) or known sensitivity to mammalian-derived products.
* Subject has plasma cell leukemia (according to World Health Organization [WHO] criterion: ≥20% of cells in the peripheral blood with an absolute plasma cell count of more than 2 × 109/L) or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
* Subject is known or suspected of not being able to comply with the study protocol (eg, because of alcoholism, drug dependency, or psychological disorder). Subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise the well-being) or that could prevent, limit, or confound the protocol specified assessments.
* Subject is a woman who is pregnant, or breast-feeding, or planning to become pregnant while enrolled in this study within 30 days after the last dose of lenalidomide or carfilzomib, or within 4 months after the last dose of isatuximab. Or, subject is a man who plans to father a child while enrolled in this study, within 4 weeks after the last dose of lenalidomide, within 90 days of the last dose of carfilzomib, or within 4 months after the last dose of isatuximab.
* Subject has had major surgery within 2 weeks before enrollment or has not fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study. Kyphoplasty or vertebroplasty is not considered major surgery.
* Subject has received an investigational drug (including investigational vaccines) or used an invasive investigational medical device within 4 weeks before enrollment or is currently enrolled in an interventional investigational study.
* Subject has contraindications to required prophylaxis for deep vein thrombosis and pulmonary embolism.
* Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs.
* Peripheral neuropathy ≥ Grade 2 on clinical examination during the screening period.
* Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobartital), or use of Ginkgo biloba, St. John's wort within 14 days before the first dose of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2022-07-30 (Actual); Study Completion 2026-03-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth O'Donnell, MD, Principal Investigator — Massachusetts General Hospital
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: MGH - Contact the Partners Innovations team at http://www.partners.org/innovation

REFERENCES:
- [Derived] O'Donnell E, Mo C, Yee AJ, Nadeem O, Laubach J, Rosenblatt J, Munshi N, Midha S, Cirstea D, Chrysafi P, Horick N, Richardson PG, Raje N. Isatuximab, carfilzomib, lenalidomide, and dexamethasone in patients with newly diagnosed, transplantation-eligible multiple myeloma (SKylaRk): a single-arm, phase 2 trial. Lancet Haematol. 2024 Jun;11(6):e415-e424. doi: 10.1016/S2352-3026(24)00070-X. Epub 2024 Apr 24. PMID 38677302

RESULTS

PARTICIPANT FLOW:
Groups:
- Induction: All participants will receive 4 cycles of induction therapy. Based on the recommendation of investigators, participants may or may not proceed to an autologous stem cell transplant (SCT) after cycles 1-4. Each cycle is 28 days in length (see dosing details below.)
  For patient undergoing upfront stem cell transplant (SCT): 4 cycles followed by stem cell collection, high-dose chemotherapy, and autologous SCT followed by 2 cycles (called consolidation).
  For patients deferring SCT following collection: 4 cycles followed by stem cell collection followed by 4 additional cycles.
  Carfilzomib: 56 mg/m2 IV on days 1, 8,15 Lenalidomide 25 mg orally (PO) on Days 1-21 Isatuximab: 10 mg/kg IV weekly for cycles 1-2 (days 1, 8, 15, 22), then every 2 weeks for cycles 3-6 (days 1 and 15), and monthly (day 1) thereafter Dexamethasone: 20 mg orally (PO) administered day of and day after carfilzomib and isatuximab (days 1, 2, 8, 9, 15, and 16; days 22 and 23 during cycles 1-2 only).
  Patients achieving a partial response (PR) or greater will be stratified by cytogenetic risk and receive either high risk (Lenalidomide 10 mg orally (PO) Day 1-21 Carfilzomib 56 mg/m2 or last tolerated dose IV Days 1, 15 Isatuximab 10 mg/kg IV Day 1) or low risk maintenance therapy (Lenalidomide 10 mg orally (PO) Day 1-21).
Period: Overall Study
Arm/Group | Induction
Started | 50
Completed | 47
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Induction
Number analyzed (Participants) | 50
Age, Continuous [Median (Full Range); unit: years] | 59 [37 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 44
  More than one race | 0
  Unknown or Not Reported | 1
ISS Stage at Diagnosis [Count of Participants; unit: Participants] — The International Staging System (ISS) for multiple myeloma predicts the severity of multiple myeloma based on routinely obtained lab values (serum beta-2 microglobulin and serum albumin), with severity increasing from Stage I to Stage III.
  Stage I: serum beta-2 microglobulin less than 3.5 mg/L and serum albumin greater than or equal to 3.5 g/dL.
  Stage II: serum beta-2 microglobulin less than 3.5 mg/L and serum albumin less than 3.5 g/dL, OR beta-2 microglobulin 3.5 to 5.5 mg/L, irrespective of serum albumin.
  Stage III: serum beta-2 microglobulin greater than 5.5 mg/L
  Participants
    I | 28
    II | 16
    III | 6
Revised ISS Stage at Diagnosis [Count of Participants; unit: Participants] — The Revised International Staging System (R-ISS) predicts the severity of myeloma, with severity increasing from Stage I to III.
  I: serum beta-2 microglobulin less than 3.5 mg/L, serum albumin greater than or equal to 3.5 g/dL, no high-risk chromosomal abnormalities (CA)* by fluorescence in-situ hybridization (FISH), normal lactate dehydrogenase (LDH)
  II: does not meet criteria for R-ISS Stage I or III.
  III: serum beta-2 microglobulin greater than or equal to than 5.5 mg/L AND high-risk CA* by FISH OR high LDH
  *High risk CAs: del(17p), translocation t(4;14), translocation t(14;16)
  Participants
    I | 16
    II | 32
    III | 2
ECOG Performance Status [Count of Participants; unit: Participants] — ECOG performance status describes a patient's level of functioning in terms of their ability to care for themself, daily activity, and physical ability.
  Grade 0: Fully active, able to carry on all pre-disease performance without restriction Grade 1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  Participants
    0 | 28
    1 | 22
High Risk Cytogenetics [Count of Participants; unit: Participants] — High risk cytogenetics defined as deletion 17p, gain of 1q, and translocations t(4:14), t(14;16), and/or t(14;20).
  Participants
    Yes | 23
    No | 23
    Unknown | 4
Serum Heavy Light Chain [Count of Participants; unit: Participants]
  IgG | 20
  IgA | 13
  Light-chain only | 10
  Unknown | 7

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR + Stringent CR) Rate
Description: Percentage of patients who achieved a complete response (CR) or stringent CR (sCR) per International Myeloma Working Group (IMWG) Uniform Response criteria after 4 cycles of of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI). IMWG criteria define a CR as "Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow" and an sCR as "CR plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence."
Time Frame: 112 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Induction
Number analyzed (Participants) | 47
Participants | 19

2. Secondary Outcome: Overall Response Rate After 4 Cycles Induction Therapy
Description: Overall response rate will be the percentage of patients who achieve at least partial response (PR) per International Myeloma Working Group (IMWG) Uniform Response criteria after 4 cycles of of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI).
  The IMWG response criteria define a PR as:
  > 50% reduction of serum M-protein and reduction in 24 hours urinary M-protein by >90% or to < 200 mg/24 h, OR If the serum and urine M-protein are unmeasurable, a > 50% decrease in the difference between involved and uninvolved FLC levels in place of the M-protein criteria, OR If serum and urine M-protein are not measurable, and serum free light assay is also not measurable, > 50% reduction in plasma cells is required in place of M-protein, provided baseline bone marrow plasma cell percentage was > 30%.
  In addition to the above listed criteria, if present at baseline, a > 50% reduction in the size of soft tissue plasmacytomas is also required for a partial response.
Time Frame: 112 days (4 cycles)
Measure: Count of Participants; unit: Participants
Arm/Group | Induction
Number analyzed (Participants) | 47
Participants | 47

3. Secondary Outcome: Minimal Residual Disease (MRD) Rate After 4 Cycles Induction Therapy
Description: MRD is the small number myeloma cells surviving in the bone marrow after a clinical response has been measured and the patient is in remission. MRD negativity will be determined by deep sequencing of genomic deoxyribonucleic acid from bone marrow samples using rearranged Ig locus-specific primers (Adaptive, Seattle, WA). The MRD rate after 4 cycles of of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI) is the percentage of patients who are MRD negative at 10^(-5) and 10^(-6), meaning that no MRD was detected in samples of 100,000 cells and 1,000,000 cells, respectively.
Time Frame: 112 Days (4 Cycles)
Population: After cycle 4, 28 patients out of 47 patients evaluable for response had evaluable MRD data.
Measure: Count of Participants; unit: Participants
Arm/Group | Induction
Number analyzed (Participants) | 28
Participants
  MRD negative at 10^(-5) | 12
  MRD negative at 10^(-6) | 9

4. Secondary Outcome: Minimal Residual Disease (MRD) Rate at 10^(-5) in Patients Receiving Upfront Stem Cell Transplant
Description: MRD is the small number myeloma cells surviving in the bone marrow after a clinical response has been measured and the patient is in remission. MRD negativity will be determined by deep sequencing of genomic deoxyribonucleic acid from bone marrow samples using rearranged Ig locus-specific primers (Adaptive, Seattle, WA). The MRD rate is the percentage of patients who are MRD negative at 10^(-5), meaning that no MRD was detected in a sample of 100,000 cells. MRD status was assessed after 4 cycles of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI) induction, stem cell transplant, and 2 cycles of KRDI consolidation therapy (6 cycles total.)
Time Frame: 168 Days (6 cycles, upfront transplant)
Population: Of all patients enrolled to the main arm of the protocol (induction), 47 were evaluable for response. Of these 47 patients, 5 received upfront stem cell transplant. All five patients receiving upfront SCT had evaluable MRD results.
Measure: Number; unit: percentage of participants
Groups:
- Upfront Stem Cell Transplant (4 Cycles Induction Therapy, SCT, and 2 Cycles Consolidation Therapy): All participants will receive 4 cycles of induction therapy. Based on the recommendation of investigators, participants may or may not proceed to an autologous stem cell transplant (SCT) after cycles 1-4. Each cycle is 28 days in length (see dosing details below.)
  For patient undergoing upfront stem cell transplant (SCT): 4 cycles followed by stem cell collection, high-dose chemotherapy, and autologous SCT followed by 2 cycles (called consolidation).
  For patients deferring SCT following collection: 4 cycles followed by stem cell collection followed by 4 additional cycles.
  Carfilzomib: 56 mg/m2 IV on days 1, 8,15 Lenalidomide 25 mg orally (PO) on Days 1-21 Isatuximab: 10 mg/kg IV weekly for cycles 1-2 (days 1, 8, 15, 22), then every 2 weeks for cycles 3-6 (days 1 and 15), and monthly (day 1) thereafter Dexamethasone: 20 mg orally (PO) administered day of and day after carfilzomib and isatuximab (days 1, 2, 8, 9, 15, and 16; days 22 and 23 during cycles 1-2 only).
  Patients achieving a partial response (PR) or greater will be stratified by cytogenetic risk and receive either high risk (Lenalidomide 10 mg orally (PO) Day 1-21 Carfilzomib 56 mg/m2 or last tolerated dose IV Days 1, 15 Isatuximab 10 mg/kg IV Day 1) or low risk maintenance therapy (Lenalidomide 10 mg orally (PO) Day 1-21).
Arm/Group | Upfront Stem Cell Transplant (4 Cycles Induction Therapy, SCT, and 2 Cycles Consolidation Therapy)
Number analyzed (Participants) | 5
percentage of participants | 20

5. Secondary Outcome: Minimal Residual Disease (MRD) Rate at 10^(-5) in Patients Deferring Stem Cell Transplant
Description: MRD is the small number myeloma cells surviving in the bone marrow after a clinical response has been measured and the patient is in remission. MRD negativity will be determined by deep sequencing of genomic deoxyribonucleic acid from bone marrow samples using rearranged Ig locus-specific primers (Adaptive, Seattle, WA). The MRD rate is the percentage of patients who are MRD negative at 10^(-5), meaning that no MRD was detected in a sample of 100,000 cells. MRD status was assessed after 4 cycles of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI) induction, stem cell collection, and 4 additional cycles of KRDI (8 cycles total).
Time Frame: 224 Days (8 cycles transplant-deferred)
Population: Of all patients enrolled to the main arm of the protocol (induction), 47 were evaluable for response. Of these 47 patients, 42 deferred stem cell transplant. 35 of these 42 patients had evaluable MRD results.
Measure: Count of Participants; unit: Participants
Groups:
- Deferred Stem Cell Transplant (4 Cycles, Stem Cell Collection, 4 Additional Cycles): All participants will receive 4 cycles of induction therapy. Based on the recommendation of investigators, participants may or may not proceed to an autologous stem cell transplant (SCT) after cycles 1-4. Each cycle is 28 days in length (see dosing details below.)
  For patient undergoing upfront stem cell transplant (SCT): 4 cycles followed by stem cell collection, high-dose chemotherapy, and autologous SCT followed by 2 cycles (called consolidation).
  For patients deferring SCT following collection: 4 cycles followed by stem cell collection followed by 4 additional cycles.
  Carfilzomib: 56 mg/m2 IV on days 1, 8,15 Lenalidomide 25 mg orally (PO) on Days 1-21 Isatuximab: 10 mg/kg IV weekly for cycles 1-2 (days 1, 8, 15, 22), then every 2 weeks for cycles 3-6 (days 1 and 15), and monthly (day 1) thereafter Dexamethasone: 20 mg orally (PO) administered day of and day after carfilzomib and isatuximab (days 1, 2, 8, 9, 15, and 16; days 22 and 23 during cycles 1-2 only).
  Patients achieving a partial response (PR) or greater will be stratified by cytogenetic risk and receive either high risk (Lenalidomide 10 mg orally (PO) Day 1-21 Carfilzomib 56 mg/m2 or last tolerated dose IV Days 1, 15 Isatuximab 10 mg/kg IV Day 1) or low risk maintenance therapy (Lenalidomide 10 mg orally (PO) Day 1-21).
Arm/Group | Deferred Stem Cell Transplant (4 Cycles, Stem Cell Collection, 4 Additional Cycles)
Number analyzed (Participants) | 35
Participants | 26

6. Secondary Outcome: Progression Free Survival at 12 Months
Description: Progression free survival (PFS) is defined as the time between the start of treatment and disease progression or death due to any cause. PFS at 12 months is the percentage of patients who were alive and without disease progression 12 months after initiating treatment with of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI).
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction
Number analyzed (Participants) | 47
percentage of participants | 97.9 [95.9 to 99.7]

7. Secondary Outcome: Overall Survival at 12 Months
Description: Overall survival (OS) is defined as the time between the start of treatment and death due to any cause. OS at 12 months is the percentage of patients who were alive 12 months after initiating treatment with of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI).
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Induction
Number analyzed (Participants) | 47
percentage of participants | 97.9 [86.1 to 99.7]

8. Secondary Outcome: Complete Response Rate in Patients With Upfront Stem Cell Transplant
Description: Percentage of patients who achieved a complete response (CR) or stringent CR (sCR) per International Myeloma Working Group (IMWG) Uniform Response criteria after 4 cycles of of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI), stem cell transplant, and 2 cycles of KRDI consolidation (6 cycles total). IMWG criteria define a CR as "Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow" and an sCR as "CR plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence."
Time Frame: 168 Days
Population: Of all patients enrolled to the main arm of the protocol (induction), 47 were evaluable for response. Of these 47 patients, 5 received upfront stem cell transplant.
Measure: Number; unit: percentage of participants
Arm/Group | Upfront Stem Cell Transplant (4 Cycles Induction Therapy, SCT, and 2 Cycles Consolidation Therapy)
Number analyzed (Participants) | 5
percentage of participants | 80

9. Secondary Outcome: Complete Response Rate in Patients Deferring Stem Cell Transplant
Description: Percentage of patients who achieved a complete response (CR) or stringent CR (sCR) per International Myeloma Working Group (IMWG) Uniform Response criteria after 4 cycles of of Isatuximab, Carfilzomib, Lenalidomide, and Dexamethasone (KRDI), stem cell collection, and 4 additional cycles of KRDI after deferring stem cell transplant (8 cycles total). IMWG criteria define a CR as "Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow" and an sCR as "CR plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence."
Time Frame: 224 Days
Population: Of all patients enrolled to the main arm of the protocol (induction), 47 were evaluable for response. Of these 47 patients, 42 deferred stem cell transplant.
Measure: Number; unit: percentage of participants
Arm/Group | Deferred Stem Cell Transplant (4 Cycles, Stem Cell Collection, 4 Additional Cycles)
Number analyzed (Participants) | 42
percentage of participants | 67

ADVERSE EVENTS:
Time Frame: The AE data reported here extends from the start of study treatment through cycle 8 (224 days).
Arm/Group | Induction
All-Cause Mortality (participants affected / at risk) | 1/50
Serious Adverse Events (participants affected / at risk) | 8/50
Other Adverse Events (participants affected / at risk) | 49/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Induction (N=50)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Spinal Fracture (Injury, poisoning and procedural complications) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary Emboli
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — COVID-19
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Non-arteritic anterior ischemic optic neuropathy (NAION)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Acute Kidney Injury (Renal and urinary disorders) | 2 (2)
Right Hip Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction (N=50)
Abdominal pain (Gastrointestinal disorders) | 3
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 24
Alkaline phosphatase increased (Investigations) | 17
Allergic Reaction (Immune system disorders) | 1
Allergic Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anemia (Blood and lymphatic system disorders) | 21
Ankle fracture (Injury, poisoning and procedural complications) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 14
Atrial fibrillation (Cardiac disorders) | 1
Autoimmune Disorder (Immune system disorders) | 1 — Rheumatoid Arthritis
Back Pain (Musculoskeletal and connective tissue disorders) | 19
Bloating (Gastrointestinal disorders) | 4
Blood bilirubin increased (Investigations) | 6
Blood lactate dehydrogenase increased (Investigations) | 10
Blurred vision (Eye disorders) | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 10
Bruising (Injury, poisoning and procedural complications) | 2
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — Chest tightness
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — Bradycardia
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — Holosystolic murmur
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — Tachycardia
Cardiac troponin T increased (Investigations) | 1
Cataract (Eye disorders) | 2
Chest pain - cardiac (Cardiac disorders) | 1 — Chest congestion
Chills (General disorders) | 5
Cholesterol high (Investigations) | 1
Chronic Kidney Disease (Renal and urinary disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Concentration impairment (Nervous system disorders) | 3
Conjunctivitis (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Creatinine increased (Investigations) | 8
Cyanosis (Cardiac disorders) | 17
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 20
Dizziness (Nervous system disorders) | 12
Dry mouth (Gastrointestinal disorders) | 5
Dysgeusia (Nervous system disorders) | 7
Dyspepsia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Edema limbs (Gastrointestinal disorders) | 14
Endocrine disorders - Other, specify (Endocrine disorders) | 1 — Decreased vitamin D level
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1 — Scratched cornea
Eye disorders - Other, specify (Eye disorders) | 1 — Stye of left eyelid
Eye disorders - Other, specify (Eye disorders) | 1 — Ocular hypertension
Eye disorders - Other, specify (Eye disorders) | 1 — Retinal hemorrhage
Eye disorders - Other, specify (Eye disorders) | 1 — Red and crusty eyes
Fatigue (General disorders) | 35
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Fever (General disorders) | 10
Flank pain (Musculoskeletal and connective tissue disorders) | 2
Flatulence (Gastrointestinal disorders) | 2
Flu like symptoms (General disorders) | 5
Flushing (Vascular disorders) | 4
Fracture, anterior ribs and wrist (Injury, poisoning and procedural complications) | 1
Gait disturbance (General disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Suspected GI bleed
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — GI Upset
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Melena s/p colonoscopy
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Soft yellow stool
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Seasonal allergies
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Head cold
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Lumps in right armpit
General disorders and administration site conditions - Other, specify (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
GGT increased (Investigations) | 1
Glucose intolerance (Metabolism and nutrition disorders) | 1
Hallucinations (Nervous system disorders) | 1
Headache (Nervous system disorders) | 15
Hearing impaired (Ear and labyrinth disorders) | 1
Hematoma (Vascular disorders) | 1
Hematuria (Renal and urinary disorders) | 2
Hemolysis (Blood and lymphatic system disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 4
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hot flashes (Vascular disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 22
Hyperkalemia (Metabolism and nutrition disorders) | 2
Hyperlipidemia (Metabolism and nutrition disorders) | 6
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 22
Hyperthyroidism (Endocrine disorders) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 8
Hypocalcemia (Metabolism and nutrition disorders) | 22
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 9
Hypophosphatemia (Metabolism and nutrition disorders) | 22
Hypotension (Vascular disorders) | 4
Hypothyroidism (Endocrine disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Infections and infestations - Other, specify (Infections and infestations) | 9 — COVID-19 infection
Infused related reaction (Injury, poisoning and procedural complications) | 10
Injection site reaction (General disorders) | 1
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 — Food poisoning
Insomnia (Psychiatric disorders) | 21
Irritability (Psychiatric disorders) | 4
Localized edema (General disorders) | 1
Viral Meningitis (Infections and infestations) | 1
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 — Diabetes
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 — Hyperbilirubinemia
Muscle cramp (Musculoskeletal and connective tissue disorders) | 7
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Pain and swelling in right foot
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Hip pain
Myalgia (Musculoskeletal and connective tissue disorders) | 6
Nail discoloration (Skin and subcutaneous tissue disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9
Nausea (Gastrointestinal disorders) | 23
Neck pain (Musculoskeletal and connective tissue disorders) | 4
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Tingling in toes
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Tastebud change
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Neuropathy
Nervous system disorders - Other, specify (Nervous system disorders) | 1
Neutrophil count decreased (Investigations) | 29
Non-cardiac chest pain (General disorders) | 6
Obesity (Metabolism and nutrition disorders) | 4
Oral pain (Gastrointestinal disorders) | 2
Pain (General disorders) | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Papulopustular rash (Infections and infestations) | 2
Paresthesia (Nervous system disorders) | 2
Paroxysmal atrial tachycardia (Cardiac disorders) | 1
Pelvic pain (Reproductive system and breast disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 2
Peripheral sensory neuropathy (Nervous system disorders) | 7
Platelet count decreased (Investigations) | 16
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 5
Psychiatric disorders - Other, specify (Psychiatric disorders) | 4 — Mood changes
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 — Bipolar disorder 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 14
Renal and urinary disorder - Other, specify (Renal and urinary disorders) | 1 — Sensation in perineum
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Asthma
Restlessness (Psychiatric disorders) | 1
Rhinitis infective (Infections and infestations) | 22
Sinus bradycardia (Cardiac disorders) | 2
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2
Sinus tachycardia (Cardiac disorders) | 3
Sinusitis (Infections and infestations) | 3
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Diaphoresis
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Scalp rash; spread to ears, chest, arms
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Small lesion on right upper cheek
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — petechiae noted on bilateral forearms
Skin infection (Infections and infestations) | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3
Spinal Fracture (Injury, poisoning and procedural complications) | 1
Stomach pain (Gastrointestinal disorders) | 1
Syncope (Nervous system disorders) | 1
Testicular disorder (Reproductive system and breast disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Thrush (Infections and infestations) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Tooth development disorder (Gastrointestinal disorders) | 1 — Broken teeth
Tooth Infection (Infections and infestations) | 1
Toothache (Gastrointestinal disorders) | 2
Tremor (Nervous system disorders) | 3
Upper respiratory infection (Infections and infestations) | 9
Urinary tract pain (Renal and urinary disorders) | 1
Urinary urgency (Renal and urinary disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Vascular disorders - Other, specify (Vascular disorders) | 1 — Increased fluid retention
Vision decreased (Eye disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight loss (Investigations) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
White blood cell decreased (Investigations) | 26
Wound complication (Injury, poisoning and procedural complications) | 2
Wrist fracture (Injury, poisoning and procedural complications) | 1

LIMITATIONS AND CAVEATS:
Results up to cycle 6/8 of KRDI are currently available and entered in CT.gov, including the primary endpoint and secondary endpoints that can be reported at this time. Data after the beginning of maintenance therapy (post-cycle 6 for patients who had stem cell transplants, and post-cycle 8 for patients who deferred stem cell transplant), including adverse event data, is still being collected and analyzed as of August 2023.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-02): https://cdn.clinicaltrials.gov/large-docs/94/NCT04430894/Prot_SAP_001.pdf
  • Informed Consent Form (2023-05-01): https://cdn.clinicaltrials.gov/large-docs/94/NCT04430894/ICF_002.pdf